CLINICAL TRIAL: NCT02970864
Title: A Phase I Trial of a Novel Synthetic Polymer Nerve Conduit 'Polynerve' in Participants With Sensory Digital Nerve Injury
Acronym: UMANC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Principal Investigator, Adam Reid, Chief Investigator, University of Manchester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R116863; 2016-001667-37 (EudraCT Number)
Record Dates: First submitted 2016-11-15; First posted 2016-11-22 (Estimated); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Injury of Nerves at Wrist and Hand Level
Keywords: Nerve regeneration; Peripheral nerve injury; Nerve conduits; Sensory nerve transection
MeSH Terms: conditions — Peripheral Nerve Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Polynerve (Experimental): Participants found to have a nerve gap of at least 5 mm and no greater than 20mm will undergo repair with the Polynerve.
  Interventions: Device: Polynerve

INTERVENTIONS:
Device: Polynerve — Polymer biomaterial nerve conduit

SUMMARY:
Participants with a traumatic sensory nerve injury in the hand will be recruited to the study. Participants found to have a nerve gap of at least 5 mm and no greater than 20mm will undergo repair with the Polynerve. Participants will be followed up regularly, observed for device-related complications and to assess the return of sensory innervation.

DETAILED DESCRIPTION:
Peripheral nerve injuries are a common occurrence, with approximately 9000 cases in the United Kingdom (UK) occurring each year. Most are in a predominantly young and working population. Where surgical reconstruction is required to repair the peripheral nerve injury, techniques employed have changed little in the last 50-60 years with many factors influencing the outcomes, such as age of patient, timing, level and extent of injury, method of repair and the surgeon's skill .

Despite advances in microsurgical nerve repair techniques, functional recovery is often poor e.g. resulting impaired hand sensation, reduced motor function and frequent pain and cold intolerance. This can have a profound and permanent impact on the patient's recovery and subsequent quality of life. Nerve repair has significant health, social and cost implications with the treatment and rehabilitation of an employed person, estimated to be EUR 51,238.

Peripheral nerve injury usually presents with nerve stumps that can be approximated in surgical repair: direct, end-to-end suture repair of the epineurium (neurorrhaphy). Excessive tension over the suture line leads to poor results; therefore when the nerve stumps cannot be approximated without tension, an alternative surgical method is required.

Where the nerve gap exceeds more than 5 mm, there are two fundamental options, either 'nerve grafting' or 'tubulisation' using a bridging material. This trial will examine the first-in-man use of a new nerve conduit device 'Polynerve' to repair small nerve gaps in digital sensory nerves of the hand. Polynerve is a degradable co-polymer of Poly ε-caprolactone (PCL) and Poly (L-lactic acid) (PLA) which is shaped as a cylinder with a novel internal lumen consisting of a specific micro-grooved architecture.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any trial specific procedures
2. Traumatic injury/injuries to the hand with clinical suspicion of sensory nerve transection mandating surgical exploration
3. Male and females aged 18-80

Exclusion Criteria:

1. Concomitant injuries requiring surgical treatment from other specialists
2. Specified co-morbidities that would increase a participants risk of infection including diabetes, renal/liver disease, autoimmune diseases, primary or secondary immunocompromised participants (including immunosuppressive drugs or known disease resulting in suppressed immunity)
3. A stated hypersensitivity or allergy to the polymers PCL/PLA
4. Any other significant co-morbidity impacting on the risk of surgery (to be determined by the multi-disciplinary team (MDT))
5. Known to have participated in a clinical trial of an investigational agent or device in the previous 30 days.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-08-17 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2021-05-06 (Actual)

PRIMARY OUTCOMES:
Assessment of safety and tolerability: number of patients with treatment-related adverse events as assessed by the Clavien-Dindo classification of surgical complications | 1 year
  To assess the safety and tolerability of use of the polymer biomaterial nerve conduit to repair a sensory nerve transection of the hand

SECONDARY OUTCOMES:
Measurement of efficacy: Sensory nerve function measured by two-point discrimination (2PD), the Weinstein Enhanced Sensory Test (WEST) monofilaments, and locognosia | 1 year
  To measure efficacy of the polymer biomaterial nerve conduit to support nerve regeneration following the transection of the sensory nerve of the hand

CONTACTS AND LOCATIONS:
Overall Officials: Adam Reid, Study Chair — University of Manchester
Locations (1):
- Wythenshawe Hospital, Manchester University NHS Foundation Trust, Wythenshawe, Manchester, United Kingdom

REFERENCES:
- [Derived] Murphy R, Faroni A, Wong J, Reid A. Protocol for a phase I trial of a novel synthetic polymer nerve conduit 'Polynerve' in participants with sensory digital nerve injury (UMANC). F1000Res. 2019 Jun 24;8:959. doi: 10.12688/f1000research.19497.1. eCollection 2019. PMID 32685131